CLINICAL TRIAL: NCT04852380
Title: Clinical Results Of Platelet Rich Plasma (PRP) Injections For Knee Osteoarthritis (KOA), Our Experience At Midterm Follow Up
Brief Title: Platelet Rich Plasma (PRP) Injections For Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Other Study IDs: PRP-Knee Osteoarthritis
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoarthritis (KOA); Platelet-rich plasma (PRP);
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated by PRP injection
  Interventions: Procedure: PRP injections

INTERVENTIONS:
Procedure: PRP injections — The 5 mL PRP concentrate was injected every week for three times, starting from recruitment. The patient was placed supine whit a knee flexion of 90°.All the procedures were carried out in an aseptic condition, injected in the knee soft spot through an anterior approach, using a 21-gauge needle.

SUMMARY:
It was conducted a prospective study with a series of 153 patients treated with PRP injections in patient affected by knee osteoarthritis. One independent observer performed clinical and functional evaluations at T0 (recruitment), T1 (one month after the injection), T2 (three months after the last injection) and T3 (six months after the last injection).

The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), the Knee Score Society (KSS) score and the Visual Analogue Scale (VAS) were evaluated and recorded for each patient at each follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age between 40 and 81;
* Body mass index (BMI) between 21.5 and 29.3;
* Chronic history (for at least 4 months) of knee joint pain;
* Radiographically documented knee osteoarthritis of grades 1 to 3 (Kellgren-Lawrence (K-L) radiographic classification scale)

Exclusion Criteria:

* Radiographically severe documented knee osteoarthritis of grade 4 (K-L radiographic classification scale);
* Previous femur and tibia fractures;
* Knee previous surgical treatment (e.g., arthroscopy);
* Hyaluronic acid infiltration within the previous six months;
* Hemoglobin levels <10 g/dL;
* History of oncohematological disease, infections, or immunodepression

Ages: 40 Years to 81 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred and fiftythree patients referring to the Orthopaedic and Trauma Unit of the local University Hospital between January 2018 and January 2020 with knee osteoarthritis
Sampling Method: Probability Sample
Enrollment: 153 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogic Scale | Day 0; Month 1; Month 3; Month 6 (after the injection)
  The knee pain was quantified using the Visual Analogic Scale ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- AOUC Policlinico di Bari - UOC Ortopedia e Traumatologia, Bari, Italy